CLINICAL TRIAL: NCT06815406
Title: Recurrence Rate After Endoscopic Resection of , Laterally Spreading Tumor Granular Type (LST-G) of the Colon and Rectum: Endoscopic Mucosal Resection (EMR) Vs. Endoscopic Submucosal Dissection (ESD): a Multicenter Randomized Controlled Trial ( ESD Vs EMR )
Brief Title: Recurrence Rate After Endoscopic Resection of , Laterally Spreading Tumor Granular Type (LST-G) of the Colon and Rectum: Endoscopic Mucosal Resection Vs. Endoscopic Submucosal Dissection
Acronym: ESD vs EMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104/2021/SPER/IRCCSRE
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
Keywords: Endoscopic Mucosal Resection (EMR); Endoscopic submucosal dissection (ESD); Laterally spreading tumors (LST)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic Mucosal Resection (EMR) (Active Comparator)
  Interventions: Procedure: Endoscopic Mucosal Resection (EMR)
- Endoscopic Submucosal Dissection (ESD) (Experimental)
  Interventions: Procedure: Endoscopic Submucosal Dissection (ESD)

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection (EMR) — atients assigned to this arm will undergo Endoscopic Mucosal Resection (EMR), a standard endoscopic technique that involves the resection of colorectal Laterally Spreading Tumors - Granular type (LST-G) using a diathermic snare with submucosal injection. The procedure may be performed en bloc or in a piecemeal fashion, depending on lesion size and characteristics. EMR is widely accepted for lesions with low submucosal invasion risk but has a higher recurrence rate than ESD.
  Arms: Endoscopic Mucosal Resection (EMR)
Procedure: Endoscopic Submucosal Dissection (ESD) — Patients assigned to this arm will undergo Endoscopic Submucosal Dissection (ESD), an advanced endoscopic technique that allows for en bloc resection of large colorectal Laterally Spreading Tumors - Granular type (LST-G). The procedure involves the use of specialized knives to dissect the submucosal layer, ensuring complete resection with histologically clear margins (R0 resection). ESD has been associated with lower recurrence rates but requires a high level of expertise, longer procedural times, and carries a higher risk of complications.
  Arms: Endoscopic Submucosal Dissection (ESD)

SUMMARY:
Colorectal cancer is one of the leading causes of cancer-related mortality worldwide. Early-stage non-polypoid neoplastic lesions, particularly Laterally Spreading Tumors - Granular Type (LST-G) larger than 20mm, require effective endoscopic removal to prevent malignant progression. The two primary techniques for resecting these lesions are Endoscopic Mucosal Resection (EMR) and Endoscopic Submucosal Dissection (ESD).

EMR is a widely used, minimally invasive technique that involves resecting the lesion with a diathermic snare after submucosal injection. While effective and safe, EMR often necessitates piecemeal resection, increasing the risk of local recurrence. In contrast, ESD, developed in Asia, allows for en bloc resection regardless of lesion size, ensuring more accurate histopathological assessment and lower recurrence rates. However, ESD requires greater technical expertise, has longer procedural times, and carries a higher risk of complications.

In Western clinical practice, EMR remains the standard treatment, whereas ESD is selectively performed in high-expertise centers. Given the lack of randomized controlled trials comparing EMR and ESD in Western populations, this study aims to provide robust clinical evidence to guide treatment decisions.

The primary objective of this study is to compare the recurrence/residual adenomatous tissue rate at 6 and 12 months between EMR and ESD in patients with LST-G lesions of the colon and rectum

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of Laterally Spreading Tumor - Granular Type (LST-G) ≥ 20 mm in the colon or rectum with an indication for endoscopic resection.
* Life expectancy > 10 years.
* Ability to understand and sign the informed consent form, demonstrating comprehension of the study and willingness to participate.

Exclusion Criteria:

* Diagnosis of Laterally Spreading Tumor - Non-Granular Type (LST-NG).
* Presence of depressed areas within the lesion.
* Lesions located on a scar or anastomosis site.
* Lesions classified as Kudo Vi or Vn pattern.
* History of chronic inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease).
* Diagnosis of hereditary polyposis syndromes (e.g., familial adenomatous polyposis, Lynch syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence/Adenomatous Residual Rate | 6 and 12 months after treatment
  Proportion of patients with local recurrence or residual adenomatous tissue, confirmed through follow-up colonoscopies and histopathological examination.

SECONDARY OUTCOMES:
Complete Resection Rate | 6 and 12 months after treatment
  Proportion of patients with a complete histopathological resection (R0), defined as tumor-free margins in both lateral and deep resection edges, out of the total number of randomized patients
Differences in Procedure Time | Up to 2 months
  Comparison of the average duration of the procedure (from submucosal injection to complete lesion resection) between the EMR and ESD groups. The procedure time is measured intraoperatively and is calculated as the total duration from the initial submucosal injection to the completion of lesion resection.
Bleeding Rate | During procedure (up to 2 months from enrollment) and 24 hours and 3 months after treatment
  Number of patients experiencing bleeding out of the total number of randomized patients.
Perforation Rate | During procedure (up to 2 months from enrollment) and 24 hours and 3 months after treatment
  Number of patients with an intraoperative perforation, defined as visible mesenteric fat or free peritoneal space during the procedure, or delayed perforation diagnosed based on symptoms (abdominal pain, fever, peritonitis) and confirmed by radiological imaging (free air, fluid collection).
Overall Complication Rate | 24 hours after treatment
  Proportion of patients experiencing at least one complication, classified according to the Accordion Severity Classification of Postoperative Complications.

CONTACTS AND LOCATIONS:
Overall Officials: Sassatelli Romano, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (5):
- Italy (5):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna - Sant'Orsola Malpighi, Bologna
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Università Vita Salute - IRCCS, Milan
  - Ospedale Civile di Baggiovara, Modena
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogie RMM, Veldman MHJ, Snijders LARS, Winkens B, Kaltenbach T, Masclee AAM, Matsuda T, Rondagh EJA, Soetikno R, Tanaka S, Chiu HM, Sanduleanu-Dascalescu S. Endoscopic subtypes of colorectal laterally spreading tumors (LSTs) and the risk of submucosal invasion: a meta-analysis. Endoscopy. 2018 Mar;50(3):263-282. doi: 10.1055/s-0043-121144. Epub 2017 Nov 27. PMID 29179230
- [Background] Kudo S, Hirota S, Nakajima T, Hosobe S, Kusaka H, Kobayashi T, Himori M, Yagyuu A. Colorectal tumours and pit pattern. J Clin Pathol. 1994 Oct;47(10):880-5. doi: 10.1136/jcp.47.10.880. PMID 7962600
- [Background] Oka S, Tanaka S, Saito Y, Iishi H, Kudo SE, Ikematsu H, Igarashi M, Saitoh Y, Inoue Y, Kobayashi K, Hisabe T, Tsuruta O, Sano Y, Yamano H, Shimizu S, Yahagi N, Watanabe T, Nakamura H, Fujii T, Ishikawa H, Sugihara K; Colorectal Endoscopic Resection Standardization Implementation Working Group of the Japanese Society for Cancer of the Colon and Rectum, Tokyo, Japan. Local recurrence after endoscopic resection for large colorectal neoplasia: a multicenter prospective study in Japan. Am J Gastroenterol. 2015 May;110(5):697-707. doi: 10.1038/ajg.2015.96. Epub 2015 Apr 7. PMID 25848926
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Fujiya M, Tanaka K, Dokoshi T, Tominaga M, Ueno N, Inaba Y, Ito T, Moriichi K, Kohgo Y. Efficacy and adverse events of EMR and endoscopic submucosal dissection for the treatment of colon neoplasms: a meta-analysis of studies comparing EMR and endoscopic submucosal dissection. Gastrointest Endosc. 2015 Mar;81(3):583-95. doi: 10.1016/j.gie.2014.07.034. Epub 2015 Jan 13. PMID 25592748
- [Background] Moss A, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Burgess NG, Sonson R, Byth K, Bourke MJ. Long-term adenoma recurrence following wide-field endoscopic mucosal resection (WF-EMR) for advanced colonic mucosal neoplasia is infrequent: results and risk factors in 1000 cases from the Australian Colonic EMR (ACE) study. Gut. 2015 Jan;64(1):57-65. doi: 10.1136/gutjnl-2013-305516. Epub 2014 Jul 1. PMID 24986245
- [Background] Pimentel-Nunes P, Dinis-Ribeiro M, Ponchon T, Repici A, Vieth M, De Ceglie A, Amato A, Berr F, Bhandari P, Bialek A, Conio M, Haringsma J, Langner C, Meisner S, Messmann H, Morino M, Neuhaus H, Piessevaux H, Rugge M, Saunders BP, Robaszkiewicz M, Seewald S, Kashin S, Dumonceau JM, Hassan C, Deprez PH. Endoscopic submucosal dissection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Sep;47(9):829-54. doi: 10.1055/s-0034-1392882. Epub 2015 Aug 28. PMID 26317585
- [Background] Tanaka S, Kashida H, Saito Y, Yahagi N, Yamano H, Saito S, Hisabe T, Yao T, Watanabe M, Yoshida M, Kudo SE, Tsuruta O, Sugihara KI, Watanabe T, Saitoh Y, Igarashi M, Toyonaga T, Ajioka Y, Ichinose M, Matsui T, Sugita A, Sugano K, Fujimoto K, Tajiri H. JGES guidelines for colorectal endoscopic submucosal dissection/endoscopic mucosal resection. Dig Endosc. 2015 May;27(4):417-434. doi: 10.1111/den.12456. Epub 2015 Mar 5. PMID 25652022
- [Background] Fuccio L, Repici A, Hassan C, Ponchon T, Bhandari P, Jover R, Triantafyllou K, Mandolesi D, Frazzoni L, Bellisario C, Bazzoli F, Sharma P, Rosch T, Rex DK. Why attempt en bloc resection of non-pedunculated colorectal adenomas? A systematic review of the prevalence of superficial submucosal invasive cancer after endoscopic submucosal dissection. Gut. 2018 Aug;67(8):1464-1474. doi: 10.1136/gutjnl-2017-315103. Epub 2017 Dec 5. PMID 29208675
- [Background] Strasberg SM, Linehan DC, Hawkins WG. The accordion severity grading system of surgical complications. Ann Surg. 2009 Aug;250(2):177-86. doi: 10.1097/SLA.0b013e3181afde41. PMID 19638919
- [Background] Yoshida M, Kakushima N, Mori K, Igarashi K, Kawata N, Tanaka M, Takizawa K, Ito S, Imai K, Hotta K, Ishiwatari H, Matsubayashi H, Ono H. Learning curve and clinical outcome of gastric endoscopic submucosal dissection performed by trainee operators. Surg Endosc. 2017 Sep;31(9):3614-3622. doi: 10.1007/s00464-016-5393-9. Epub 2016 Dec 30. PMID 28039646